CLINICAL TRIAL: NCT00803816
Title: Everolimus for the Treatment of Uveitis Unresponsive to Cyclosporine A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carsten Heinz (Other)
Responsible Party: Sponsor-Investigator, Carsten Heinz, Prof Heiligenhaus Head of Department, St. Franziskus Hospital
Organization: St. Franziskus Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-004876-10
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Uveitis
Keywords: endogoneous; posterior; intermediate
MeSH Terms: conditions — Uveitis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Addition of everolimus to standard care (Other): refractive to cyclosporine A (CsA) received additional everolimus.
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — everolimus 1.0 - 2.5mg oral daily dosage

SUMMARY:
Study efficacy of everolimus on course of uveitis:

* obtain quiescence of inflammation after start of treatment
* duration to obtain quiescence of inflammation
* number of patients with quiescence of inflammation

DETAILED DESCRIPTION:
occurence of new complications from uveitis

* course of visual acuity (LogMAR): percentage of patients with visual loss of 10 or more numbers on ETDRS as compared to baseline
* change of recurrence rate as compared to time before everolimus treatment
* occurence of recurrence after obtaining remission with everolimus treatment
* duration to occurence of recurrence o number of patients with recurrence
* corticosparing effect from everolimus
* number of patients without topical corticosteroids; number of patients with reduced topical corticosteroids (<3x/daily)
* number of patients without systemic corticosteroids; number of patients with reduced systemic corticosteroids (<10mg/daily)
* efficacy of uveitis within 12 months
* maintenance of remission after withdrawel of everolimus treatment at 12 months o course of cystoid macula edema (FLA, OCT)

ELIGIBILITY:
Inclusion Criteria:

* endogenous intermediate or posterior uveitis
* no quiesence in previous 3 months under systemic and topical steroids or systemic cyclosporine A
* indication for steroid sparing therapy
* uveitis related vision threating complications
* negative pregnancy test
* effective contraception

Exclusion Criteria:

Ophthalmic parameters:

* silicone oil in anterior chamber of both eyes para- or intraocular corticosteroid injections within previous 8 weeks
* opacities of optic media that obscure visualization of anterior or posterior eye segments

General parameters:

* requirement for combined immunosuppression for systemic immune-mediated disease contraindication against everolimus or cyclosporine A
* positive tuberculine test (GT 10
* currently immunosuppressive therapy with immunosuppressive drug other than cyclosporine
* poor compliance
* known intolerance to medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Inactivity of uveitis | 1 year

SECONDARY OUTCOMES:
Reoccurence of uveitis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Heiligenhaus, MD, Principal Investigator — Department of Ophthalmology at St. Franziskus Hospital
Locations (1):
- Department of Ophthalmology at St. Franziskus Hospital, Münster, Germany